CLINICAL TRIAL: NCT04286555
Title: Dietary Approaches to Stop Hypertension for Diabetes Trial
Brief Title: Dietary Approaches to Stop Hypertension for Diabetes
Acronym: DASH4D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Sheikh Khalifa Stroke Institute at Johns Hopkins (Unknown); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00232059; R01DK128900 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes; Diabetes type2; Type2 Diabetes; Type 2 Diabetes; Type II Diabetes; Hypertension; High Blood Pressure
Keywords: diet; DASH; sodium
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Intervention Model Description: The study design is a four-period crossover feeding study, in which participants will be randomly assigned to an order of four isocaloric diets for a 5-week period each.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators and the outcomes assessors will not know which order of diets the participant has been assigned. The participant will not be explicitly told which diet he or she is receiving during each period, but by the nature of higher sodium vs. lower sodium or the differences between the DASH4D and comparison diet, the participant would likely be able to guess based on the menus and taste.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DASH4D diet with lower sodium (Active Comparator): DASH-style dietary pattern, modified for people with diabetes, with sodium level of 1500 mg/day
  Interventions: Other: DASH4D diet; Other: lower sodium
- DASH4D diet with higher sodium (Active Comparator): DASH-style dietary pattern, modified for people with diabetes, with sodium level of 3700 mg/day
  Interventions: Other: DASH4D diet; Other: higher sodium
- Comparison diet with lower sodium (Active Comparator): Dietary pattern that is typical of what many Americans with diabetes eat, with sodium level of 1500 mg/day
  Interventions: Other: comparison diet; Other: lower sodium
- Comparison diet with higher sodium (Other): Dietary pattern that is typical of what many Americans with diabetes eat, with sodium level of 3700 mg/day
  Interventions: Other: comparison diet; Other: higher sodium

INTERVENTIONS:
Other: DASH4D diet — DASH stands for "Dietary Approaches to Stop Hypertension". The DASH diet is a healthy dieter that lowers blood pressure. The DASH diet emphasizes fruits, vegetables, and low-fat dairy products; includes whole grains, poultry, fish, and nuts; and is reduced in red meat, sweets, and sugar-containing beverages. The DASH4D dietary pattern is a version of the DASH diet that is lower in carbohydrate.
  Arms: DASH4D diet with higher sodium; DASH4D diet with lower sodium
Other: comparison diet — The comparison dietary pattern is based on a typical American diet, with macronutrient distributions generally at the average of typical US intake, and micronutrient targets generally near the 25th percentile of usual US intake (with the exception of sodium).
  Arms: Comparison diet with higher sodium; Comparison diet with lower sodium
Other: higher sodium — 3700 mg/day sodium (at the 2000 kilocalorie level)
  Arms: Comparison diet with higher sodium; DASH4D diet with higher sodium
Other: lower sodium — 1500 mg/day sodium (at the 2000 kilocalorie level)
  Arms: Comparison diet with lower sodium; DASH4D diet with lower sodium

SUMMARY:
The objective of the DASH4D trial is to determine the effects, alone and combined, of (a) the DASH4D diet (a DASH-style diet modified for people with diabetes) vs. comparison diet that is typical of what many Americans with diabetes eat and (b) lower sodium intake vs. higher sodium intake on blood pressure (BP). The core design is a single-site, 4-period, crossover feeding study with 5-week periods. Participants are fed each of four isocaloric diets, presented in random order. The primary contrast of interest is DASH4D diet with lower sodium vs. comparison diet with higher sodium.

DETAILED DESCRIPTION:
DASH4D Main Trial:

In persons with and without diabetes, elevated blood pressure (BP) is the leading cause of stroke and a major risk factor for other cardiovascular diseases, including coronary heart disease and heart failure. Strategies that effectively lower BP include drug therapy and lifestyle modification. Lifestyle modifications, particularly dietary approaches, have been shown to lower BP in persons without diabetes. However, there is a striking dearth of evidence on BP-lowering, lifestyle modifications, other than weight loss, in persons with diabetes. The DASH4D trial is designed to provide this evidence.

The DASH4D trial builds upon the investigators' experience in four NIH-sponsored feeding studies (DASH, DASH-Sodium, OmniHeart, and OmniCarb). The trial will enroll approximately 100 adults with Type 2 diabetes, systolic BP 120-159 mmHg, and diastolic BP <100 mmHg, to determine the effects, alone and combined, of (a) the DASH4D diet (a DASH-style diet modified for people with diabetes) vs. comparison diet (typical of what many Americans with diabetes eat) and (b) lower sodium intake vs. higher sodium intake on BP.

The core design is a four-period, single-site, crossover feeding study with 5-week periods. Participants are fed each of four diets, presented in random order:

1. DASH4D diet with lower sodium
2. DASH4D diet with higher sodium
3. comparison diet with lower sodium
4. comparison diet with higher sodium.

The primary contrast of interest is the DASH4D diet with lower sodium vs. the comparison diet with higher sodium.

The DASH4D diet is similar to the original DASH diet, but is lower in carbohydrates and higher in unsaturated fat than the original DASH diet, and therefore, is more consistent with dietary recommendations for persons with diabetes than the original DASH diet. The comparison diet reflects what many persons with diabetes currently consume. The lower sodium intake of approximately 1500 mg/day (at 2000 kcal) has been shown to lower BP in persons without diabetes, and has been recommended in some dietary guidelines. The higher sodium intake of approximately 3700 mg/day (at 2000 kcal) is based on estimated average intake in the US.

Outcomes are measured at the end of each feeding period. The primary outcome is end-of-period, office-based systolic BP. Other outcomes are diastolic BP, measures of glycemia, plasma lipid risk factors, patient symptoms, and estimated cardiovascular disease risk.

Similar to the investigators' prior feeding studies, the investigators expect that the results of the DASH4D trial will be immediately applicable to public health and clinical guidelines and will influence nutrition policy. Furthermore, the trial will provide a rigorous platform to assess the impact of diet and sodium intake on a diverse array of other outcomes in persons with Type 2 diabetes.

DASH4D CONTINUOUS GLUCOSE MONITORING (CGM) ANCILLARY STUDY:

Continuous glucose monitoring (CGM) systems are novel technologies recommended for assessing real-time glucose patterns, biochemical hypoglycemia, and glycemic variability. The DASH4D-CGM ancillary study will offer CGM to all participants in the DASH4D trial during a screening visit and during the two weeks at the end of each of four feeding periods.

CGM outcomes will be based on CGM data captured from week 3 to week 5 (up to 14 days) of each 5-week feeding period. Per current analytic recommendations, CGM outcomes will be generated using all available CGM data for each feeding period. The primary CGM outcomes are mean glucose, time-in-range (percentage of time glucose is between 70 and 180 mg/dL), and coefficient of variation. These outcomes were selected based on clinical guidelines and recommendations from a consensus statement on CGM endpoints for clinical trials.

We hypothesized that salt would have no effect on glucose. Therefore, we plan to combine data from the lower and higher sodium feeding periods for each diet to increase statistical power. Our primary aim is to examine the average difference in mean glucose, time-in-range, and coefficient of variation between the DASH4D and comparison diets.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 or older
* Diabetes Mellitus Type 2 defined by HbA1c ≥6.5% or treatment of diabetes with diabetes medication(s)
* Baseline systolic BP of 120-159 mmHg (based on average across 3 screening visits)
* Baseline diastolic BP <100 mmHg (based on average across 3 screening visits)
* Willing and able to eat on site for one meal per day, 3 days per week, and eat only and all food provided as part of the study diets during the controlled feeding periods (run-in and four 5-week feeding periods). Note that actual frequency of on-site dining may be fewer than 3 days per week due to COVID-related restrictions, but participants will still need to be on site to pick up food and be weighed 3 days per week, and will still be expected to have meals monitored (in-person or remotely) for one meal per day, 3 days per week.
* Willing and able to complete required measurement procedures
* Have access to a mobile device or computer with video conference capabilities, or be willing to use a device for video conferencing provided by the study

EXCLUSION CRITERIA:

* Laboratory Exclusions

  * Serum potassium ≥5.2 mmol/L or <3.5 mmol/L
  * Estimated glomerular filtration rate (eGFR) <30 mL/min by commercial lab result (note that prior to 7/12/22, the lab was using the race-based Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation, and on/after 7/12/22, the lab switched to using the CKD-EPI 2021 equation, which does not provide different estimated GFR by race))
  * HbA1c>9.0%
* Medication Exclusions

  1. Unstable dose (i.e., change in the 2 months prior to screening or prior to randomization) of any of the following:

     * Anti-hypertensive medications
     * Sodium-glucose co-transporter 2 (SGLT2) inhibitors or glucagon-like peptide-1 (GLP-1) receptor agonists
     * Stimulants, including oral medications for asthma or chronic obstructive pulmonary disease (COPD)
     * Hormone replacement therapy or thyroid hormone
     * Weight-increasing psychotropic agents, including antipsychotic agents, lithium, and mirtazapine
  2. Use of any of the following medications:

     * Potassium supplementation in any form, including a multivitamin or electrolyte drink mix, with a dose >99 mg/day, which is the allowable amount in over-the-counter products
     * Prandial or short-acting insulin
     * GLP-1 receptor agonist if on weight loss dose
     * Warfarin (Coumadin)
     * Chronic oral corticosteroid (intermittent use is okay)
     * Weight loss medications
     * Tirzepatide (Mounjaro)
  3. Unwillingness to keep same dose of vitamin, mineral, and botanical supplements
  4. Any medication not compatible with participation as determined by the investigators
* Medical History Exclusions

  * Type 1 diabetes
  * Hypoglycemia requiring hospitalization or the assistance of another person in the last 12 months
  * Active cardiovascular disease or any event in the prior 6 months, including coronary artery bypass grafting (CABG), percutaneous transluminal coronary angioplasty (PTCA), myocardial infarction (MI), cerebrovascular accident (CVA), or congestive heart failure (CHF) exacerbation requiring hospital admission
  * Cancer diagnosis or treatment in the last 2 years (benign tumors or non-melanoma skin cancer or localized breast or prostate cancer not requiring chemotherapy is acceptable)
  * Active inflammatory bowel disease, bowel resection, malabsorptive syndrome, pancreatitis (episode within past year), history of Roux-en-Y gastric bypass, or history of other bariatric surgery that limits food intake volume or that requires a specific diet plan
  * Pregnancy or lactation or planned pregnancy
  * Any emergency department (ED) visit for asthma or chronic obstructive pulmonary disease (COPD) in the last 6 months
  * Any other serious illness or condition not compatible with participation as determined by the investigators
* Physical Exclusions

  * Body weight >420 pounds
  * Arm circumference ≥50cm
  * Weight loss or gain of >5.0% of body weight during 2 months prior to screening, or large weight change during screening prior to randomization
* Lifestyle and Other Exclusions

  * Significant food allergies, preferences, intolerances, or dietary requirements that would interfere with diet adherence
  * Not able to self-monitor glucose if needed
  * Consumption of more than 14 alcoholic drinks per week or consumption of more than 6 drinks on one or more occasion per week
  * Active substance use disorder that would interfere with participation
  * Participation in or planning to start weight loss program
  * Current participation in another clinical trial that might affect blood pressure or ability to comply with study procedures
  * Planning to leave area prior to end of study
  * Investigator discretion

DASH4D-CGM ANCILLARY STUDY EXCLUSION CRITERIA:

All DASH4D main trial participants will be invited to participate in the embedded CGM ancillary study. Participants with the following contraindications to wearing a CGM sensor will be excluded from the ancillary study:

* History of allergic skin reaction to adhesive
* Implantable pacemaker

Note: Participants excluded from, or who do not wish to participate in, the CGM ancillary study are still allowed to participate in the DASH4D main trial if eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2024-06-13 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (SBP) | At the end of 5-week feeding period
  After the participant has rested quietly in the seated position for at least 5 minutes, blood pressure will be measured in triplicate, using an Omron device, with each reading separated by 30 seconds, and the average of the three readings (in mmHg) will also be recorded. Blood pressure will be measured on five separate occasions during the last 2 weeks of the feeding period, and the mean systolic blood pressure from these five blood pressures (15 total readings) will be used as the primary outcome.

SECONDARY OUTCOMES:
Diastolic blood pressure (DBP) | At the end of 5-week feeding period
  After the participant has rested quietly in the seated position for at least 5 minutes, blood pressure will be measured in triplicate, using an Omron device, with each reading separated by 30 seconds, and the average of the three readings (in mmHg) will also be recorded. Blood pressure will be measured on five separate occasions during the last 2 weeks of the feeding period, and the mean diastolic blood pressure from these five blood pressures (15 total readings) will be used as a secondary outcome.

OTHER OUTCOMES:
Glycated albumin level | At the end of 5-week feeding period
  Glycated albumin percentage (%).
Fructosamine level | At the end of 5-week feeding period
  Fructosamine level in mmol/L.
Fasting glucose level | At the end of 5-week feeding period
  Fasting glucose level in mg/dL.
Hemoglobin A1c (HbA1c) level | At the end of 5-week feeding period
  HbA1c percentage (%).
Cardiovascular disease (CVD) risk percentage | At the end of 5-week feeding period
  Current 10-year atherosclerotic cardiovascular disease (ASCVD) risk will be reported as a percent, using the American College of Cardiology (ACC)/American Heart Association (AHA) ASCVD risk equation.
Total cholesterol level | At the end of 5-week feeding period
  Total cholesterol level in mg/dL.
Low-density lipoprotein (LDL) cholesterol level | At the end of 5-week feeding period
  LDL cholesterol level in mg/dL.
High-density lipoprotein (HDL) cholesterol level | At the end of 5-week feeding period
  HDL cholesterol level in mg/dL.
Triglyceride level | At the end of 5-week feeding period
  Triglyceride level in mg/dL.
Presence of orthostatic hypotension | At the end of 5-week feeding period
  Participants will lie in the supine position for 5 minutes and undergo three blood pressure measurements, separated by 30 seconds. The average of these three readings will be used as the supine blood pressure. Participants will stand with their arm rested on an adjacent Mayo table at 70-80 degrees from their torso, and participants will then undergo another set of triplicate blood pressure measurements, separated by 30 seconds each. The average of these three readings will be used as the standing blood pressure. Presence of orthostatic hypotension will be defined as ≥ 20 mmHg drop in systolic blood pressure or a ≥ 10 mmHg drop in diastolic blood pressure upon standing.
Postural change in systolic blood pressure | At the end of 5-week feeding period
  Participants will lie in the supine position for 5 minutes and undergo three blood pressure measurements, separated by 30 seconds. The average of these three readings will be used as the supine blood pressure. Participants will stand with their arm rested on an adjacent Mayo table at 70-80 degrees from their torso, and participants will then undergo another set of triplicate blood pressure measurements, separated by 30 seconds each. The average of these three readings will be used as the standing blood pressure. Change in systolic blood pressure (mmHg) upon standing will be calculated.
Postural change in diastolic blood pressure | At the end of 5-week feeding period
  Participants will lie in the supine position for 5 minutes and undergo three blood pressure measurements, separated by 30 seconds. The average of these three readings will be used as the supine blood pressure. Participants will stand with their arm rested on an adjacent Mayo table at 70-80 degrees from their torso, and participants will then undergo another set of triplicate blood pressure measurements, separated by 30 seconds each. The average of these three readings will be used as the standing blood pressure. Change in diastolic blood pressure (mmHg) upon standing will be calculated.
Symptoms experienced by participants as assessed by a questionnaire | At the end of 5-week feeding period
  Participants will complete a questionnaire about symptoms experienced while on each diet, including symptoms related to fall risk (e.g., feeling faint), food intake and output (e.g., bloating, constipation), fluid intake and output (e.g., excessive thirst), and general symptoms (e.g., fatigue or low energy). Participants will be asked to rate each listed symptom as: did not occur, mild, moderate, or severe. Score range 0-69, higher score worse symptoms.
Mean continuous glucose monitoring sensor glucose | At the end of 5-week feeding period
  CGM Ancillary Study Primary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The mean of these glucose measurements (in mg/dL) during the 14-day wear period will be used as a primary outcome of the corresponding feeding period.
Percentage of time glucose between 70 and 180 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Primary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was between 70 and 180 mg/dL (time-in-range) during 14-day wear period will be used as a primary outcome of the corresponding feeding period.
Glucose coefficient of variation (%) | At the end of 5-week feeding period
  CGM Ancillary Study Primary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The glucose coefficient of variation (standard deviation divided by mean glucose, multiplied by 100 and expressed as a percent) during the 14-day wear period will be used as a primary outcome of the corresponding feeding period.
Glucose standard deviation | At the end of 5-week feeding period
  CGM Ancillary Study Secondary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The standard deviation of glucose measurements (in mg/dL) will be used as a secondary outcome of the corresponding feeding period.
Percentage of time glucose above 180 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Secondary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was above 180 mg/dL during the 14-day wear period will be used as a secondary outcome of the corresponding feeding period.
Percentage of time glucose above 250 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Secondary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was above 250 mg/dL during the 14-day wear period will be used as a secondary outcome of the corresponding feeding period.
Percentage of time glucose below 70 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Secondary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was below 70 mg/dL during the 14-day wear period will be used as a secondary outcome of the corresponding feeding period.
Percentage of time glucose below 54 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Secondary Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was below 54 mg/dL during the 14-day wear period will be used as a secondary outcome of the corresponding feeding period.
Percentage of time glucose between 70 to 140 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was between 70 and 140 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Percentage of time glucose above 140 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The percentage of time glucose was above 140 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with >70% time glucose between 70 to 180 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants that spent >70% of time with glucose between 70 and 180 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with glucose coefficient of variation <36% | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants with a glucose coefficient of variation <36% during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with <25% time glucose above 180 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants that spent <25% of time with glucose above 180 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with <5% time glucose above 250 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants that spent <5% of time with glucose above 250 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with <4% time glucose below 70 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants that spent <4% of time with glucose below 70 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.
Proportion of participants with <1% time glucose below 54 mg/dL | At the end of 5-week feeding period
  CGM Ancillary Study Other Outcome: Continuous glucose monitoring sensors will be worn up to 14 days during each 5-week feeding period in participants included in the DASH4D-CGM ancillary study. The proportion of participants that spent <1% of time with glucose below 54 mg/dL during the 14-day wear period will be used as an exploratory outcome of the corresponding feeding period.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appel, MD, MPH, Principal Investigator — Johns Hopkins University; Hsin Chieh Yeh, PhD, Principal Investigator — Johns Hopkins University; Scott Pilla, MD, MHS, Principal Investigator — Johns Hopkins University; Elizabeth Selvin, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins ProHealth, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fang M, Wang D, Rebholz CM, Echouffo-Tcheugui JB, Tang O, Wang NY, Mitchell CM, Pilla SJ, Appel LJ, Selvin E. DASH4D diet for glycemic control and glucose variability in type 2 diabetes: a randomized crossover trial. Nat Med. 2025 Oct;31(10):3309-3316. doi: 10.1038/s41591-025-03823-3. Epub 2025 Aug 5. PMID 40764427
- [Derived] Pilla SJ, Yeh HC, Mitchell CM, Miller ER 3rd, Oh S, White K, Durkin N, Stein AA, Charleston JB, Lu M, Hu X, Wu B, Selvin E, Fang M, Maruthur NM, Juraschek SP, Mueller NT, Wang NY, Appel LJ; DASH4D Collaborative Research Group. Dietary Patterns, Sodium Reduction, and Blood Pressure in Type 2 Diabetes: The DASH4D Randomized Clinical Trial. JAMA Intern Med. 2025 Aug 1;185(8):937-946. doi: 10.1001/jamainternmed.2025.1580. PMID 40489102